CLINICAL TRIAL: NCT04846894
Title: Diagnostic Performance of Ga-68 PSMA-11 PET/CT in Patients With Biochemical Recurrence After Prostatectomy: A Comparison of Digital PET/CT and Analog PET/CT Scanner Images
Brief Title: Ga-68 PSMA-11 PET/CT in Patients With Biochemical Recurrence of Prostate Cancer: Digital PET/CT Versus Analog PET/CT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jin-Sook Ryu (Other)
Responsible Party: Sponsor-Investigator, Jin-Sook Ryu, Professor, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AMC 2021-0195
Record Dates: First submitted 2021-04-13; First posted 2021-04-15 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Biochemical Recurrence; Ga-68 PSMA-11 PET/CT
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biochemical Recurrence (Experimental): Prostate cancer patient with biochemical recurrence
  Interventions: Diagnostic Test: Ga-68 PSMA-11 PET/CT imaging

INTERVENTIONS:
Diagnostic Test: Ga-68 PSMA-11 PET/CT imaging — Sequential PET/CT imaging using analog and digital PET/CT scanners after single intravenous injection of Ga-68 PSMA-11

SUMMARY:
Ga-68 PSMA-11 PET/CT is known as useful method for localizing recurred tumor lesions in prostate cancer patients with biochemical recurrence [elevated serum prostate specific antigen (PSA) after radical prostatectomy]. The recent digital PET/CT which is known to show better resolution and sensitivity than analogue PET/CT may have better performance for detecting early small recurred tumor lesions. This study is intended to compare the diagnostic performance (detection rate and positive predictive value) of Ga-68 PSMA-11 PET/CT using analogue PET/CT scanner and digital PET/CT scanner in same patients who had biochemical recurrence of prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Preliminary study - Establishment of Ga-68 PSMA-11 PET/CT imaging conditions (three subjects)

   * Equal or more than 19 years old
   * Biopsy proven prostate cancer patients with high risk group (serum PSA> 20 ng/ml) or metastatic prostate cancer patients identified on other imaging modalities prior to Ga-68 PSMA-11 PET/CT imaging
2. Main study (40 subjects)

   * Equal or more than 19 years old
   * Patients who had previously undergone radical prostatectomy and were histologically diagnosed with prostate cancer.
   * Patients identified with biochemical recurrence through serum PSA tests during postoperative follow-up (Serum PSA level equal or more than 0.2 ng/ml at least two times and one of the tests was conducted within one month before consent to the study) in which metastatic lesions were not found or uncertain in standard imaging modalities (abdominal/Pelvic CT, bone scan).
   * Patients who can be followed up clinically, including serum PSA tests, for at least 6 months after consent to the study at this hospital.

Exclusion Criteria:

1. Preliminary study - Establishment of Ga-68 PSMA-11 PET/CT imaging conditions (three subjects)

   * Primary cancer other than prostate cancer has been previously diagnosed or has occurred simultaneously with prostate cancer; Previous primary cancer other than prostate cancer is a local disease and has been cured completely shall be an exception.
   * Subjects who has concurrent severe and/or uncontrolled and/or unstable medical disease (e.g. congestive heart failure, acute myocardial infarction, severe pulmonary disease, chronic renal or hepatic disease which could compromise participation in the study) based on the judgment of the investigator
   * Subjects who cannot perform PET/CT imaging due to claustrophobia, dyskinesia, anxiety disorders, etc.
2. Main study (40 subjects)

   * Primary cancer other than prostate cancer has been previously diagnosed or has occurred simultaneously with prostate cancer; Previous primary cancer other than prostate cancer is a local disease and has been cured completely shall be an exception.
   * Subjects who cannot perform CT, bone scan, etc., which are standard diagnostic procedures for lesion localization in case of biochemical recurrence.
   * Subjects who has concurrent severe and/or uncontrolled and/or unstable medical disease (e.g. congestive heart failure, acute myocardial infarction, severe pulmonary disease, chronic renal or hepatic disease which could compromise participation in the study) based on the judgment of the investigator
   * Subjects who cannot perform PET/CT imaging due to claustrophobia, dyskinesia, anxiety disorders, etc.
   * Subjects who might make the collection of complete data difficult or impossible due to personal circumstances or other reasons, in the judgment of the investigator.

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Detection rate and positive predictive value of Ga-68 PSMA-11 PET/CT images of digital PET/CT and analogue PET/CT | 12 months
  Comparison of detection rate and positive predictive value of Ga-68 PSMA-11 PET/CT images of digital PET/CT and analogue PET/CT in biochemical recurrence (BCR) patients

SECONDARY OUTCOMES:
Detection rate and positive predictive value of Ga-68 PSMA-11 digital and analog PET/CT according to PSA level groups | 12 months
  Comparison of detection rate and positive predictive value of Ga-68 PSMA-11 digital and analog PET/CT according to PSA level groups in BCR patients
Comparison of SUVs of Ga-68 PSMA-11 digital and analog PET/CT | 12 months
  Comparison of standardized uptake values (SUVs) of Ga-68 PSMA-11 digital and analog PET/CT

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Sook Ryu, MD.PhD., Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Songpa-gu, South Korea

IPD SHARING:
Plan to Share IPD: No